## ADAPTATION OF COMMUNITY REINFORCEMENT APPROACH FOR THE TREATMENT OF DRUG ADDICTION



**MUHAMMAD SAGHIR** 

DR. MAZHAR IQBAL BHATTI

74-FSS/PHDPSY/F-18

Associate Professor (supervisor)

**Department of Psychology** 

**Faculty of Social Sciences** 

**International Islamic University Islamabad** 

July 10, 2024

## **Background of the study**

The aim of the present study was to adapt the CRA Islamically because it is very important to add the cultural and religious aspects which are fundamentally important for the treatment of SUD. In CRA, face to face interaction is required for intervention including eight sessions for focuses on the reality of client's social environment so that for learning real life opportunities could be focused as per client needs to enhance engagement and learning (Godley, 2001).

For internal motivation and involvement in CRA, adaptations were added to enhance CRA's effectiveness. There were two major adaptations in CRA to make it accord with the cultural relevant with the targeted population. First adaptation is based on religion Islam. It includes several sections, and these sections are adapted in CRA's counseling goals. In first section morality was adapted with CRA, morality is about the Islamically integrated ways about hygiene, sleep, eating, clothes, meeting others, physical health, happiness and sadness related (Abbass, 2017). Second section was related to internal framework of human psyche, which comprises of Cognition (Aql), Behavioral inclinations (Nafs), Spirit (Ruh), Emotions (Ihsaas) and Heart (Qalb) (Keshavarzi & Khan, 2018). In third section principle of change, behavioral modification and tazkia-e-nafs were added along with three stages in principle of change: Inkishaf, itidal and Itehad (Keshavarzi & Khan, 2018).

## **Objectives:**

- To investigate whether IICRA has the better efficacy in treating substance dependence along with comorbidities than the indoor conventional treatment for substance dependence.
- To adapt the IICRA treatment strategy grounded in Pakistani culture and religious values for the treatment of drug addicts in Pakistan.

- To determine whether IICRA treatment is more effective in treating poly drug addicts and drug addicts with or without comorbidities.
- To determine whether IICRA treatment is more effective for those addicts who were treated for one or more treatment previously as compare to those having first treatment.

## **Research Method and Design:**

A randomized control trial was used as research method on indoor residential patients and guidelines of good clinical practices were followed (Guideline, 2001). The sample size for this clinical trial was 60 in total (30 for control group and 30 for treatment group) in order to maintain this number, the sample size was extended to 34 for each group in order to get adequate retention of the sample. The retention number of sample was 68 at the time of pre assessment and closed at 59 at the time of last follow up assessment. All participants who were admitted for treatment of SUD with or without comorbid mental disorders were recruited for research. Intervention was administered after the 21 days of detoxification. For recruitment and randomization, it was not applicable to control extraneous variables in a single facility so two sites were selected for this purpose. Selection of sites were based on minimizing extraneous variables by selecting identical residential treatment sites. One site such as Islamabad Rehab Clinic (IRC) was willing to give permission for implementation of IICRA based intervention. Hence, IRC was selected for recruiting treatment group.

Second site was considered for recruiting control group where they were giving traditional treatment in residential setting based on disease model. The site is named as Hayat Rehab Clinic (HRC). The permission for conducting research and recruiting participants were sought out from the authorities. Traditional treatment was termed as treatment as usual which includes detoxification of drugs and duration of detoxification from acute withdrawal consisted on 21 days,

during these early days focus was on adjustment to residential treatment along with hygiene and routine related compliance. Afterwards, the focus was on general counselling for drug addiction prevention, twelve steps program, habit formation based on seven habits for highly effective people and life skills training which is mainly delivered through group classes and lectures. Patients' individual sessions are also scheduled with psychologists once weekly, the focus of these individual sessions is to maximized the interaction with family through relationship building and relapse prevention skills. Duration of residential treatment is between 90-120 days.

The treatment group received interventions based on Islamically Integrated CRA (IICRA). These sessions were divided into daily goals including counseling related to hygiene, physical activities, psychotherapy of mental disorders and drug addiction related management. After discharge from residential treatment, they were followed up for six months to check the effectiveness of IICRA in the context of relapse and recovery from SUD as well as from comorbidities. These six months follow up was consist of further three follow up sessions; first session was conducted on the discharge date from the facility, second was on fifth month and third was on sixth month following discharge.

Sample in the present study for clinical trial was based on those diagnosed individuals who were hospitalized in rehab for the treatment of SUD. Age of the sample was varying from 16 years to 60 years, where 24% individuals were from late adolescence, 39% from early adulthood and finally 37% were from middle adulthood. The chronicity of disease in the sample varies 78% of them were abusing substance between from one year to 10 years and 22% were abusing more than 10 years. Similarly, the rate of relapse or number of treatments within sample was computed as 54% individuals were hospitalized first time and 46% were hospitalized two and more than two times. Additionally, the type of substance abuse was also varying cross the

sample which included cannabis, alcohol, pills, heroin, Ice and multiple substance abuse (Alcohol, cannabis and prescribed substances) as well. The gender was mainly male in sample which was 98% and only one participant was female in the sample. Moreover, 75% individuals of the sample were diagnosed with SUDs and 25% were also having comorbid mental illness. Hence, the representativeness of the sample was limited to clinical population diagnosed with SUDs as well as comorbidities with SUDs.

Secondly, the professionals who were providing treatment were not aware of the allocation of the individual in control and treatment group as well as the recruited individuals for the clinical trial. They were responsible for conducting sessions and recording those sessions through treatment forms as well as monitoring the goals whether desired goal is achieved or not. They were also given the treatment protocol schedule for effective treatment adherence.

Additionally, panel assessments were planned at both sites for reviewing and addressing treatment related issues faced by professionals as well as the achievement of desired goals of the treatment. These panel assessments were carried out by weekly to ensure the engagement of the patients, adherence and fidelity to the treatment protocols. This committee was comprised of four professionals having experience in the treatment planning and execution with the minimum educational level of MS in Clinical Psychology.

Moreover, for the purpose of comparability of results and to control the extraneous variables, two treatment sites were selected for clinical trial. Both sites were equal in terms of organizational structure which includes residential treatment facility for mental health, same geographical region with outdoor areas, hierarchy of professionals, daily routine of the patients, psychiatrist consultation, outdoor and indoor activities of the patients and length of residential

treatment. The professionals engaged in the clinical trial has similar qualification and experience at both facilities.

During this clinical trial, 28 out of 34 participants were retained in control group and successfully completed the duration of clinical trial. Three participants had withdrawn the treatment after 40 days of hospitalization and one individual passed away after discharge from rehab. Remaining two participants did not continue the follow up sessions.

Similarly, in experimental group 31 participants out of 34 had successfully completed the Treatment duration for clinical trial. Two participants had withdrawn the treatment after a month of admission and one participant did not continue after the discharge from the facility.